CLINICAL TRIAL: NCT04481035
Title: Antioxidant Therapy With N-acetylcysteine for Learning and Motor Behavior in Children With Neurofibromatosis Type 1
Acronym: NF1NAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-0344
Record Dates: First submitted 2020-04-14; First posted 2020-07-22 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-02

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Acetylcysteine; Inhalation

STUDY DESIGN:
Intervention Model Description: This is a double-blind placebo controlled, prospective, Phase IIa study to explore safety, tolerability, and efficacy of NAC on learning and motor behavior in children with NF1 aged 8 through 16 years old.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to treatment I or II (double blind: NAC study drug or placebo) for 8 weeks then cross over to the other treatment option. Drug/placebo is formulated by the investigational pharmacy at Cincinnati Children's hospital. Encapsulated drug/placebo appear identical. If drug/placebo is administered as a powder, a flavor masking agent is applied to both to enforce the participant treatment blinding. Unmasking of the treatment blind will only occur after data is collected and analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine (Experimental): Participants will be dosed with 70 mg/kg/dose (max dose 900 mg) three times per day of N-Acetylcysteine (NAC) for eight (8) weeks. This is a double-blind study, neither study participant nor study team members will know whether the participant is given study drug or placebo until after all data is collected.
  Interventions: Drug: N-acetylcysteine (NAC)
- Placebo (Placebo Comparator): Participants will be dosed three times per day with a placebo for eight (8) weeks. This is a double-blind study, neither study participant nor study team members will know whether the participant is given study drug or placebo until after all data is collected.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — The study design is essentially a cross-sectional survey and then longitudinal evaluation of cognition and behavior, motor function, cortical function, and metabolomics profiles in NF1 before and after 8 weeks of treatment with an FDA approved medication, N-acetylcysteine (NAC) or placebo. This is a cross-over double-blind placebo controlled study. Participants in the experimental phase/arm will receive 70 mg/kg/dose (max dose 900 mg) three times per day of NAC for eight (8) weeks.
  Other Names: Chemical Name: Cysteine, N-acetyl-, L; Commercial Name(s): Acetein; Acetadote, Acetylcysteine; Airbron; Broncholysin; Fluimucetin; Fluimucil; Inspir; Mucofilin; Mucomyst; Mucosolvin; NAC; Paravolex; Respaire; Synonym:L-alpha-acetamido-beta-mercaptopropionic acid; Mercapturic acid; N-Acetyl-3-mercaptoalanine; N-Acetylcysteine
  Arms: N-Acetylcysteine
Other: Placebo — The study design is essentially a cross-sectional survey and then longitudinal evaluation of cognition and behavior, motor function, cortical function, and metabolomics profiles in NF1 before and after 8 weeks of treatment with an FDA approved medication, N-acetylcysteine (NAC) or placebo. This is a cross-over double-blind placebo controlled study. Participants in the placebo phase/arm will receive placebo (non-drug) three times per day for eight (8) weeks.
  Arms: Placebo

SUMMARY:
Children with neurofibromatosis type 1 (NF1) commonly suffer from the effects of cognitive, behavioral, and motor impairments. At present there is no specific treatment for this NF1 complication. However, data from rodent models of NF1 along with uncontrolled clinical observations in children with NF1 suggest that the anti-oxidant, glutamate modulating compound N-Acetyl Cysteine (NAC) may reduce these impairments. Of particular interest is a murine study analyzing the central nervous system manifestations of NF1 at our institution. That study revealed a role for myelin-forming oligodendrocytes in the control of nitric oxide synthases (NOS) and their product, nitric oxide, in maintenance of brain structure and function, including regulation of behavior and motor control. Treating these mice with NAC corrected cellular and behavioral abnormalities. N-Acetyl Cysteine is available over the counter and has been used by thousands of individuals; moreover, it has shown some promise in clinical trials for psychiatric disorders.

In order to better understand treatment mechanisms, and possibly predict long-term outcomes, the investigators propose concurrently to explore Specific Aim 1 (1.1, 1.2, and 1.3) exploratory potential disease biomarkers as outlined below. The primary outcome of this study is motor function rated with the Physical and Neurological Examination for Subtle Signs (PANESS), a validated scale that consistently demonstrates significant impairments in children with Attention Deficit Hyperactivity Disorder (ADHD), and which our preliminary data suggest may demonstrate more extreme problems in children with NF1. The first exploratory biomarker is motor system inhibitory physiology, measured using Transcranial Magnetic Stimulation (TMS). Preliminary measures in our NF1 population also show abnormalities similar to established findings in ADHD. The second exploratory biomarker is metabolomics profiling for the biomarker of oligodendrocyte dysfunction in NF1 participants: autotaxin. Preliminary data in our NF1 population showed specific signal abnormalities in the NF1 population compared to healthy controls. Therefore, the investigators propose to perform a double-blind placebo controlled, prospective, Phase IIa study to explore safety, tolerability, and efficacy of NAC on learning and motor behavior in children with NF1 aged 8 through 16 years old.

DETAILED DESCRIPTION:
The aims of this application are to gain information in children with NF1 about possible clinical benefit of anti-oxidant treatment and to develop and evaluate quantitative brain-based and blood biomarkers relating to presence of NF1, symptom severity, and response to antioxidant therapy. Clinically, 50% of children with NF1 are underperforming or failing at school [1]. This frequently leads to decreased educational attainment and fewer opportunities as adults. An important first step was preliminary work using the PANESS scale and Transcranial Magnetic Stimulation (TMS)-evoked Short Interval Cortical Inhibition (rSICI) in children with NF1. The investigators propose to develop and extend our understanding of NF1-related motor and learning behavior in response to antioxidant therapy with NAC. The purpose of the present study is to 1) evaluate tolerability, safety, and clinical benefit of NAC in this double-blind placebo controlled study; 2) to evaluate motor function (PANESS) and physiology (TMS) biomarkers at baseline and after treatment; and 3) to quantify metabolomics profiles at baseline and after treatment. The investigators propose to study 20 children with NF1, ages 8-16 years, at baseline and after completion of 8 weeks of treatment with NAC.

NAC therapy, if successful, is expected improve these parameters. The trial endpoints are: Does behavior improve? Does motor function improve? Are there TMS biomarkers that reflect the presence of NF1 and the response to NAC treatment? Are there metabolomics measures that reflect the presence of NF1 and the response to treatment? The investigators hypothesize that predictive measures exist and can be used as a foundation for an application for funding for a larger, more definitive, placebo-controlled trial involving biomarkers and clinical outcomes. The investigators believe this work has the potential to lay groundwork for future use of relevant biomarkers for treatment and outcomes research for NF1 as well as other biologically similar conditions, collectively designated the "RASopathies" (due to involvement of the RAS family of proteins) and ultimately to guide development of more effective treatments based on disease pathophysiology.

SPECIFIC AIMS

This study involves the following aims:

Specific Aim 1: Primary Outcome of Study In children and adolescents with NF1, to characterize the behavioral and motor effects of 8 weeks of N-acetylcysteine (NAC) treatment in a cohort of 20 children and adolescents with NF1. The investigators will evaluate tolerability, safety, and clinical benefit of NAC in this double-blind crossover placebo controlled study. Aim 1.1: Characterize effects of NAC treatment on motor function in kids with NF1 using the Physical and Neurological Examination for Subtle Signs (PANESS). This is a validated scale that consistently demonstrates significant impairments in children with ADHD, and which preliminary data suggest may demonstrate more extreme problems in children with NF1 than age-matched healthy controls (unpublished data from CCHMC). The investigators hypothesize that motor function scores rated with the PANESS scale will improve after treatment with NAC. Aim 1.2: Characterize effects of NAC treatment on ADHD symptoms in children with NF1. The investigators hypothesize that ADHD attention and hyperactive/impulsive symptoms, rated with the DuPaul Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-5) based clinical rating scales, will improve after treatment with NAC.

Specific Aim 2: Experimental aim # 1 In the same cohort, the investigators will identify potential novel biomarkers of neurodevelopmental burden in NF1. Aim 2.1: Describe the function and physiology of the motor system using Transcranial Magnetic Stimulation (TMS) as a possible disease biomarker of NF1. Preliminary measures in our NF1 population also show abnormalities similar to established findings in ADHD. The investigators hypothesize that children with NF1 will have significantly less motor cortex inhibition using TMS measurements, and these measures will improve ("normalize") upon NAC treatment. The investigators will compare to age-matched healthy controls at Cincinnati Children's. Aim 2.2: The investigators propose to evaluate autotaxin as a candidate biomarker of oligodendrocyte dysfunction in NF1 participants. Preliminary data from biomarker discovery analysis of serum samples from healthy controls and NF1 patients showed lysophosphatidylcholine (LPC) depletion compared to healthy age/sex matched controls. In gene expression analysis autotaxin was elevated 4 times in neurofibroma Schwann cells compared to normal nerve Schwann cells. The investigators will collect serum and plasma from participants to assess autotaxin/LPC axis prior and post-NAC therapy. The investigators hypothesize that autotaxin axis abnormalities will be a biomarker of response to antioxidant therapy in our NF1 population.

Specific Aim 3: Experimental aim # 2 In the same cohort, to evaluate metabolomics profiles as a possible disease biomarker that is affected by NF1 and by treatment with NAC as per Aim 1. Hypothesis 4: The investigators hypothesize that specific profiles will predict clinical response to antioxidant therapy compared to age-matched healthy control (unpublished data from CCHMC).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 8 - 16 years at time of enrollment whom meet NIH diagnostic criteria for NF1.
2. Participants must have a full-scale intelligence quotient (IQ) of 70 or above, as determined by neurocognitive testing within the last 3 years or during the enrollment process.
3. Participants on stimulant or any other psychotropic medication should stay on a stable dose for at least 30 days before entering the study.

Exclusion Criteria:

1. Participants should not be receiving chemotherapy currently, or have received chemotherapy in the 6 months prior to entering the study.
2. No active intracranial lesions (stable low grade glioma are acceptable) or epilepsy diagnosis.
3. Major Depression, Bipolar Disorder, Conduct Disorder, Adjustment Disorder, other major Anxiety Disorders, or other developmental psychiatric diagnoses, based on the child's history or on parent and child responses from the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS). Note that while this is an exclusion for participation in the study if there is a prior evaluation available, this becomes a criterion, after inclusion, for the investigator to withdraw the child from the study prior to completion if identified on the first study day.
4. For females, pregnancy.
5. Current use of antidepressants, non-stimulant ADHD medications, dopamine blocking agents, mood stabilizers.
6. Implanted brain stimulator, vagal nerve stimulator, ventriculoperitoneal (VP) shunt, cardiac pacemaker, or implanted medication port.
7. Asthma (bronchospasm has been reported as occurring infrequently and unpredictable when acetylcysteine is used as a mucolytica agent).
8. High risk of upper gastrointestinal (GI) hemorrhage. Examples: presence of esophageal varices or peptic ulcers

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Gilbert, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Identifiable individual participant data will not be available to other researchers.

REFERENCES:
- [Background] Acosta MT, Gioia GA, Silva AJ. Neurofibromatosis type 1: new insights into neurocognitive issues. Curr Neurol Neurosci Rep. 2006 Mar;6(2):136-43. doi: 10.1007/s11910-996-0036-5. PMID 16522267
- [Background] Ballester R, Marchuk D, Boguski M, Saulino A, Letcher R, Wigler M, Collins F. The NF1 locus encodes a protein functionally related to mammalian GAP and yeast IRA proteins. Cell. 1990 Nov 16;63(4):851-9. doi: 10.1016/0092-8674(90)90151-4. PMID 2121371
- [Background] Rosser TL, Packer RJ. Neurocognitive dysfunction in children with neurofibromatosis type 1. Curr Neurol Neurosci Rep. 2003 Mar;3(2):129-36. doi: 10.1007/s11910-003-0064-3. PMID 12583841
- [Background] Casnar CL, Janke KM, van der Fluit F, Brei NG, Klein-Tasman BP. Relations between fine motor skill and parental report of attention in young children with neurofibromatosis type 1. J Clin Exp Neuropsychol. 2014;36(9):930-43. doi: 10.1080/13803395.2014.957166. Epub 2014 Oct 6. PMID 25284746
- [Background] Walsh KS, Janusz J, Wolters PL, Martin S, Klein-Tasman BP, Toledo-Tamula MA, Thompson HL, Payne JM, Hardy KK, de Blank P, Semerjian C, Gray LS, Solomon SE, Ullrich N; REiNS International Collaboration. Neurocognitive outcomes in neurofibromatosis clinical trials: Recommendations for the domain of attention. Neurology. 2016 Aug 16;87(7 Suppl 1):S21-30. doi: 10.1212/WNL.0000000000002928. PMID 27527646
- [Background] Acosta MT, Bearden CE, Castellanos FX, Cutting L, Elgersma Y, Gioia G, Gutmann DH, Lee YS, Legius E, Muenke M, North K, Parada LF, Ratner N, Hunter-Schaedle K, Silva AJ. The Learning Disabilities Network (LeaDNet): using neurofibromatosis type 1 (NF1) as a paradigm for translational research. Am J Med Genet A. 2012 Sep;158A(9):2225-32. doi: 10.1002/ajmg.a.35535. Epub 2012 Jul 20. PMID 22821737
- [Background] Pride N, Payne JM, Webster R, Shores EA, Rae C, North KN. Corpus callosum morphology and its relationship to cognitive function in neurofibromatosis type 1. J Child Neurol. 2010 Jul;25(7):834-41. doi: 10.1177/0883073809350723. Epub 2010 Feb 8. PMID 20142468
- [Background] Wang Y, Kim E, Wang X, Novitch BG, Yoshikawa K, Chang LS, Zhu Y. ERK inhibition rescues defects in fate specification of Nf1-deficient neural progenitors and brain abnormalities. Cell. 2012 Aug 17;150(4):816-30. doi: 10.1016/j.cell.2012.06.034. PMID 22901811
- [Background] Karlsgodt KH, Rosser T, Lutkenhoff ES, Cannon TD, Silva A, Bearden CE. Alterations in white matter microstructure in neurofibromatosis-1. PLoS One. 2012;7(10):e47854. doi: 10.1371/journal.pone.0047854. Epub 2012 Oct 19. PMID 23094098
- [Background] Gilbert DL, Isaacs KM, Augusta M, Macneil LK, Mostofsky SH. Motor cortex inhibition: a marker of ADHD behavior and motor development in children. Neurology. 2011 Feb 15;76(7):615-21. doi: 10.1212/WNL.0b013e31820c2ebd. PMID 21321335
- [Background] Chen TH, Wu SW, Welge JA, Dixon SG, Shahana N, Huddleston DA, Sarvis AR, Sallee FR, Gilbert DL. Reduced short interval cortical inhibition correlates with atomoxetine response in children with attention-deficit hyperactivity disorder (ADHD). J Child Neurol. 2014 Dec;29(12):1672-9. doi: 10.1177/0883073813513333. Epub 2014 Jan 10. PMID 24413361
- [Background] Dennis J, White MA, Forrest AD, Yuelling LM, Nogaroli L, Afshari FS, Fox MA, Fuss B. Phosphodiesterase-Ialpha/autotaxin's MORFO domain regulates oligodendroglial process network formation and focal adhesion organization. Mol Cell Neurosci. 2008 Feb;37(2):412-24. doi: 10.1016/j.mcn.2007.10.018. Epub 2007 Nov 12. PMID 18164210
- [Background] Tokumura A, Majima E, Kariya Y, Tominaga K, Kogure K, Yasuda K, Fukuzawa K. Identification of human plasma lysophospholipase D, a lysophosphatidic acid-producing enzyme, as autotaxin, a multifunctional phosphodiesterase. J Biol Chem. 2002 Oct 18;277(42):39436-42. doi: 10.1074/jbc.M205623200. Epub 2002 Aug 9. PMID 12176993
- [Background] Fox MA, Colello RJ, Macklin WB, Fuss B. Phosphodiesterase-Ialpha/autotaxin: a counteradhesive protein expressed by oligodendrocytes during onset of myelination. Mol Cell Neurosci. 2003 Jul;23(3):507-19. doi: 10.1016/s1044-7431(03)00073-3. PMID 12837632
- [Background] Chen YW, Lin HC, Ng MC, Hsiao YH, Wang CC, Gean PW, Chen PS. Activation of mGluR2/3 underlies the effects of N-acetylcystein on amygdala-associated autism-like phenotypes in a valproate-induced rat model of autism. Front Behav Neurosci. 2014 Jun 17;8:219. doi: 10.3389/fnbeh.2014.00219. eCollection 2014. PMID 24987341
- [Background] Mayes DA, Rizvi TA, Titus-Mitchell H, Oberst R, Ciraolo GM, Vorhees CV, Robinson AP, Miller SD, Cancelas JA, Stemmer-Rachamimov AO, Ratner N. Nf1 loss and Ras hyperactivation in oligodendrocytes induce NOS-driven defects in myelin and vasculature. Cell Rep. 2013 Sep 26;4(6):1197-212. doi: 10.1016/j.celrep.2013.08.011. Epub 2013 Sep 12. PMID 24035394
- [Background] Garcia RJ, Francis L, Dawood M, Lai ZW, Faraone SV, Perl A. Attention deficit and hyperactivity disorder scores are elevated and respond to N-acetylcysteine treatment in patients with systemic lupus erythematosus. Arthritis Rheum. 2013 May;65(5):1313-8. doi: 10.1002/art.37893. PMID 23400548
- [Background] Fernandes BS, Dean OM, Dodd S, Malhi GS, Berk M. N-Acetylcysteine in depressive symptoms and functionality: a systematic review and meta-analysis. J Clin Psychiatry. 2016 Apr;77(4):e457-66. doi: 10.4088/JCP.15r09984. PMID 27137430
- [Background] Hardan AY, Fung LK, Libove RA, Obukhanych TV, Nair S, Herzenberg LA, Frazier TW, Tirouvanziam R. A randomized controlled pilot trial of oral N-acetylcysteine in children with autism. Biol Psychiatry. 2012 Jun 1;71(11):956-61. doi: 10.1016/j.biopsych.2012.01.014. Epub 2012 Feb 18. PMID 22342106
- [Background] Berk M, Dean O, Cotton SM, Gama CS, Kapczinski F, Fernandes BS, Kohlmann K, Jeavons S, Hewitt K, Allwang C, Cobb H, Bush AI, Schapkaitz I, Dodd S, Malhi GS. The efficacy of N-acetylcysteine as an adjunctive treatment in bipolar depression: an open label trial. J Affect Disord. 2011 Dec;135(1-3):389-94. doi: 10.1016/j.jad.2011.06.005. Epub 2011 Jun 29. PMID 21719110
- [Background] Fluvoxamine for the treatment of anxiety disorders in children and adolescents. The Research Unit on Pediatric Psychopharmacology Anxiety Study Group. N Engl J Med. 2001 Apr 26;344(17):1279-85. doi: 10.1056/NEJM200104263441703. PMID 11323729
- [Background] Axelrod BN. Validity of the Wechsler abbreviated scale of intelligence and other very short forms of estimating intellectual functioning. Assessment. 2002 Mar;9(1):17-23. doi: 10.1177/1073191102009001003. PMID 11911230
- [Background] Zhu J, Tulsky DS, Price L, Chen HY. WAIS-III reliability data for clinical groups. J Int Neuropsychol Soc. 2001 Nov;7(7):862-6. PMID 11771629
- [Background] Mills KR, Nithi KA. Corticomotor threshold to magnetic stimulation: normal values and repeatability. Muscle Nerve. 1997 May;20(5):570-6. doi: 10.1002/(sici)1097-4598(199705)20:53.0.co;2-6. PMID 9140363
- [Background] Ziemann U. Intracortical inhibition and facilitation in the conventional paired TMS paradigm. Electroencephalogr Clin Neurophysiol Suppl. 1999;51:127-36. No abstract available. PMID 10590943
- [Background] Erkan E, Zhao X, Setchell K, Devarajan P. Distinct urinary lipid profile in children with focal segmental glomerulosclerosis. Pediatr Nephrol. 2016 Apr;31(4):581-8. doi: 10.1007/s00467-015-3239-7. Epub 2015 Nov 4. PMID 26537928
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057

RESULTS

PARTICIPANT FLOW:
Groups:
- N-Acetylcysteine Followed by Placebo: Participants will be dosed with 70 mg/kg/dose (max dose 900 mg) three times per day of N-Acetylcysteine (NAC) for eight (8) weeks, followed by placebo three times per day for 8 weeks.
- Placebo Followed by N-Acetylcysteine: Participants will be dosed three times per day with a placebo for eight (8) weeks followed by 70 mg/kg/dose (max dose 900 mg) three times per day of N-Acetylcysteine for 8 weeks.
Period: Period 1
Arm/Group | N-Acetylcysteine Followed by Placebo | Placebo Followed by N-Acetylcysteine
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Period 2
Arm/Group | N-Acetylcysteine Followed by Placebo | Placebo Followed by N-Acetylcysteine
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine Followed by Placebo | Placebo Followed by N-Acetylcysteine | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Median (Full Range); unit: years] | 13 [12 to 15] | 14.5 [12 to 17] | 13 [12 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Physical and Neurological Examination for Subtle Signs (PANESS) Total [Mean (Standard Deviation); unit: units on a scale] — Physical and Neurological Examination for Subtle Signs (PANESS) measure of motor function. The PANESS test measures timed movements, lateral preference, motor overflow, dysrhythmia, coordination, gait, balance, and motor persistence. The range of this scale is 0-119, higher scores correlate with symptom severity (worse outcome).
  units on a scale | 45 (11) | 38 (4.2) | 42 (8.7)
Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS), DuPaul DSM-5 based scale [Mean (Standard Deviation); unit: units on a scale] — Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS), DuPaul DSM-5 based clinical rating scale. The range of this scale is 0-56, higher scores correlate with symptom severity (worse outcome).
  units on a scale | 35 (5.4) | 51 (0) | 39 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Motor Function Measured by Physical and Neurological Examination for Subtle Signs (PANESS)
Description: Characterize effects of NAC treatment on motor function in kids with NF1 using the Physical and Neurological Examination for Subtle Signs (PANESS). This is a validated scale that consistently demonstrates significant impairments in children with ADHD, and which preliminary data suggest may demonstrate more extreme problems in children with NF1 than age-matched healthy controls (unpublished data from CCHMC). The investigators hypothesize that motor function scores rated with the PANESS scale will improve after treatment with NAC. The range of this scale is 0-119, higher scores correlate with symptom severity (worse outcome).
Time Frame: At baseline and end of 8 weeks treatment with either NAC or placebo (weeks 0 and 8 for treatment phase one of this cross-over double blind study and at weeks 10 and 18 for treatment phase two).
Population: Descriptive only
Measure: Median (Full Range); unit: score on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale | 0 [-8 to 2] | 3 [-4 to 25]

2. Primary Outcome: Change From Baseline in ADHD Symptoms as Reported Via Parent/Teacher Surveys
Description: Characterize effects of NAC treatment on ADHD symptoms in children with NF1. The investigators hypothesize that ADHD attention and hyperactive/impulsive symptoms, rated with the DuPaul DSM-5 based clinical rating scales, will improve after treatment with NAC. The range of this scale is 0-56, higher scores correlate with symptom severity (worse outcome).
Time Frame: as for outcome 1
Population: Modified ITT - all participants who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -12.5 (13.1) | -3.75 (12.0)

3. Secondary Outcome: Transcranial Magnetic Stimulation (TMS) - Cortical Silent Period
Description: Transcranial Magnetic Stimulation (TMS) - Cortical Silent Period (CSP). This measure describes the function and physiology of the motor system using Transcranial Magnetic Stimulation (TMS) over the brain to evoke a muscle twitch in the hand. These evoked potentials provide information about the instantaneous balance of excitation and inhibition in the brain, which in turn relate in part to neurotransmitter levels that can be altered by diseases and by treatments. This measure reflects an inhibitory neurotransmitter called GABA-B and its action at a particular receptor - the "GABA B" receptor. A lengthening of the duration of CSP indicates more inhibition, which is good (within a healthy range of approximately 50 to 150 ms, because outside of that range is abnormal). Here we report the average difference before and after treatment.
Time Frame: as for outcome 1
Population: modified ITT - at least one dose given
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 5 | 5
ms | 6 (19) | -4 (18)

4. Secondary Outcome: Metabolic Testing Biomarkers
Description: The investigators propose to evaluate the autotaxin/LPC axis. High autotaxin levels correlate with a worse outcome. Low lysophosphatidylcholine (LPC) levels correlate to a worse outcome. The investigators will collect serum and plasma from participants to assess autotaxin/LPC axis prior and post-NAC therapy.
  We will perform serum targeted analysis for LPC, autotaxin activity and LPA measurements pre and post-treatment. We will perform a highly specific mass spectrometry target analysis of LPC species from serum for clinical correlation. We will use authentic standards to accurately measure low and high levels of these biomarkers. We will quantify autotaxin enzyme activity using a fluorometric assay to correlate with LPC measurements. We will quantify LPA using serum ELISA kit.
  Data is not yet available as the samples in storage for follow up study.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2025-12

5. Other Pre Specified Outcome: Evaluation of Change From Baseline in Metabolomics Profiles as a Possible Disease Biomarker Metabolic Testing Biomarkers - Samples in Storage for Follow up Study
Description: In the same cohort, to evaluate metabolomics profiles as a possible disease biomarker that is affected by NF1 and by treatment with NAC as per Aim 1. Hypothesis 4: The investigators hypothesize that specific profiles will predict clinical response to antioxidant therapy compared to age-matched healthy control (unpublished data from CCHMC).
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: 18 weeks
Groups:
- N-Acetylcysteine Treatment: Participants will be dosed with 70 mg/kg/dose (max dose 900 mg) three times per day of N-Acetylcysteine (NAC) for eight (8) weeks.
- Placebo: Participants will be dosed three times per day with a placebo for eight (8) weeks.
Arm/Group | N-Acetylcysteine Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04481035/Prot_SAP_000.pdf